CLINICAL TRIAL: NCT04667988
Title: JAK2 Mutation May Predict Response and Guide First Line Treatment in Rheumatoid Arthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: Single | Purpose: Other
Other Study IDs: R.20.11.1075
Record Dates: First submitted 2020-12-09; First posted 2020-12-16 (Actual); Last update posted 2020-12-16 (Actual); Status verified 2020-01

CONDITIONS: Response Assessment in Newly Diagnosed RA Patients at 3rd Month Was Evaluated by DAS28 and ACR in Relation to JAK Expression

STUDY DESIGN:
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- RA patients (Experimental): newly diagnosed RA will started therapy with conventional synthetic DMARDs (including methotrexate)
  Interventions: Diagnostic Test: JAK expression
- control (Experimental): JAK2 mutation assesment by PCR
  Interventions: Diagnostic Test: JAK expression

INTERVENTIONS:
Diagnostic Test: JAK expression — JAK2 assessment in blood by PCR

SUMMARY:
This study included 76 newly diagnosed RA patients and 50 matched controls. Basal JAK2 mutation was assessed by PCR in blood samples, TNF-α and IL 6 were measured by ELISA in serum of patients and controls. All patients started therapy with conventional synthetic DMARDs (including methotrexate). Response assessment at 3rd month was evaluated by DAS28 and ACR response criteria. JAK2 mutation was correlated with different clinical and laboratory parameters of patients.

DETAILED DESCRIPTION:
PCR detection of the JAK-2 V617F mutation using ASO specific PCR Genetic marker:

The detection of jak2 V617F mutation were done by using the following primers (JAK2 Reverse: 5' CTGAATAGTCCTACAGTGTTTTCAGTTTCA 3', JAK2 Forward (specific): 5' AGCATTTGGTTTTAAATTATGGAGTATATT 3' and JAK2 Forward (internal control): 5' ATCTATAGTCATGCTGAAAGTAGGAGAAAG 3'). Cycling conditions were 35 cycles with annealing temperature 58.5oC flowed by agarose gel 2% electrophoresis for bands detections.

All patients started treatment by conventional synthetic DMARDs (including methotrexate). Response assessment at 3rd month was evaluated by DAS28 and ACR response criteria. JAK2 mutation was correlated with different clinical and laboratory parameters of patients.

The Disease Activity Score (DAS) and the DAS28 have been developed to measure disease activity in RA both in daily clinical practice as well as in clinical trials on a group as well as individual level. The DAS/DAS28 is a continuous measure of RA disease activity that combines information from swollen joints, tender joints, acute phase response and general health The DAS28 is a measure of disease activity in rheumatoid arthritis (RA). DAS stands for 'disease activity score' and the number 28 refers to the 28 joints that are examined in this assessment. questionnaires (e.g. the HAQ which assesses function), X-rays, and newer imaging techniques such as ultrasound and MRI.

The ACR20 is a composite measure defined as both improvement of 20% in the number of tender and number of swollen joints, and a 20% improvement in three of the following five criteria: patient global assessment, physician global assessment, functional ability measure [most often Health Assessment Questionnaire (HAQ)], visual analog pain scale, and erythrocyte sedimentation rate or C-reactive protein (CRP). ACR50 and ACR70 are the same instruments with improvement levels defined as 50% and 70% respectively versus 20% for ACR20.

ELIGIBILITY:
Inclusion Criteria:

* New case RA patients
* good liver and renal function

Exclusion Criteria:

* Other autoimmune diss
* Malignancy
* Active viral infection
* pregnancy and lactation

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2020-04-01 (Actual); Study Completion 2020-05-01 (Actual)

PRIMARY OUTCOMES:
JAK2 mutation expression in newly diagnosed RA patients | 6 months
  Impact of pretreatment JAK2 mutation on response of Rheumatoid Arthritis patients to first line csDMARDS.

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed Elbaiomy, MD, Study Chair — Mansoura University Hospital
Locations (1):
- Mansoura University Hospital, Al Mansurah, Egypt

IPD SHARING:
Plan to Share IPD: No
Asses response of treatment in RA patients in relation to JAK2 mutation